CLINICAL TRIAL: NCT00642226
Title: A Randomized Study Comparing Combined Vitrectomy and Triamcinolone to Laser Grid in Patients With Macular Edema Secondary to Branch Retinal Vein Occlusion (BRVO)
Brief Title: Combined Vitrectomy and Triamcinolone in Macular Edema Secondary to Branch Retinal Vein Occlusion (BRVO)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to recruiting problems and the introduction of new treatment strategies (ranibizumab and dexamethasone implant).
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3.2006.1159(REK); 3.2006.1159 (Other: REK Vest, Norway); 14836 (Other: NSD, Norway)
Record Dates: First submitted 2008-03-19; First posted 2008-03-24 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Branch Retinal Vein Occlusion; Macular Edema
Keywords: Branch Retinal Vein Occlusion; BRVO; Macular Edema; Triamcinolone; Vitrectomy
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Vitrectomy; Triamcinolone; Predictive Value of Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Grid Laser
  Interventions: Procedure: Grid Laser
- 2 (Experimental): Vitrectomy in combination with 20 mg triamcinolone
  Interventions: Procedure: Vitrectomy and 20 mg triamcinolone

INTERVENTIONS:
Procedure: Grid Laser — ETDRS Grid Laser
  Other Names: Laser photocoagulation of macular edema
  Arms: 1
Procedure: Vitrectomy and 20 mg triamcinolone — Pars plana vitrectomy is followed by an injection of 20 mg purified triamcinolone acetate
  Other Names: PPV with induction of posterior vitreous detachment
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether pars plana vitrectomy in combination with triamcinolone acetate is effective in the treatment of macular edema due to branch retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Macular edema secondary to BRVO
* Best Corrected Visual Acuity of ≤ 20/40 on ETDRS chart
* Duration no shorter than 3 months
* Duration no longer than 12 months

Exclusion Criteria:

* Proliferations in study eye
* Blod in vitreous cavity
* Previous fundus laser treatment
* BRVO with over 180˚ of ischemia on FA
* Age under 18
* Other eye condition which contribute to relevant loss of visual acuity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Visual acuity (ETDRS) | 12 and 36 Months

SECONDARY OUTCOMES:
Retinal thickening measured on OCT. | 12 and 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Johan Seland, PhD, Study Director — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Department of Ophthalmology, Stavanger, Norway